CLINICAL TRIAL: NCT05318794
Title: Neoadjuvant Systemic and Peritoneal Chemotherapy for Regionally Advanced Gastric Cancer With Minimal Peritoneal Disease
Brief Title: Neoadjuvant Systemic and Peritoneal Chemotherapy for Advanced Gastric Cancer
Acronym: SPECTRA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 313621
Record Dates: First submitted 2022-03-17; First posted 2022-04-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer; Peritoneal Metastases; Chemotherapy Effect
Keywords: Pressurised intraperitoneal aerosol chemotherapy; PIPAC; Neoadjuvant therapy; Gastrectomy; Curative; Doxorubicin; Cisplatin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Doxorubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant systemic and peritoneal chemotherapy (Experimental): Standard neoadjuvant systemic and pressurised intraperitoneal aerosol chemotherapy
  Interventions: Drug: Doxorubicin and Cisplatin

INTERVENTIONS:
Drug: Doxorubicin and Cisplatin — Pressurised intraperitoneal aerosol chemotherapy
  Other Names: Adriamycin

SUMMARY:
Data demonstrating the efficacy of PIPAC in patients with regionally advanced gastric cancer with positive peritoneal cytology and/or minimal peritoneal disease is limited due to the relatively recent development of this technique and its historical preferential use in palliative patients with disseminated peritoneal metastasis.

Existing data suggest PIPAC administered every six weeks in conjunction with standard treatment may work as an adjunct to conventional systemic neoadjuvant chemotherapy. PIPAC protocols have been established both for gastric cancer as well as other intra-abdominal malignancies and have a good safety profile.

Given these promising findings, a study protocol is proposed herein to further investigate PIPAC for the treatment of a highly selected group of patients with regionally advanced gastric cancer (positive peritoneal cytology and/or minimal peritoneal disease).

DETAILED DESCRIPTION:
BACKGROUND:

There remains therefore an important, and as yet unmet, clinic need to improve survival of patients with regionally advanced gastric cancer with positive peritoneal cytology and/or minimal peritoneal disease.

To address this challenge, there has been emerging interest in the use of intraperitoneal chemotherapy for the treatment and suppression of peritoneal disease in patients with regionally advance gastric cancer.

HYPOTHESIS:

Use of combined neoadjuvant systemic chemotherapy and PIPAC in a highly selected group of patients with locally advanced gastric cancer (positive cytology and/or minimal peritoneal disease) is safe and will effectively eradicate all traces of peritoneal metastasis.

STUDY DESIGN:

This will be a non-randomised interventional cohort study of patients with regionally advanced gastric cancer (Tx, Nx) with either positive peritoneal cytology and/or minimal peritoneal disease (peritoneal carcinomatosis index, PCI ≤ 3). All patients will undergo complete cancer staging, including laparoscopy.

Prior to enrolment Potentially eligible patient will be reviewed by the Northwest London Upper Gastrointestinal Cancer Multidisciplinary Team. Study recruitment will also be open to eligible patients referred from other regional cancer networks within England. Study recruitment will also be open to eligible patients referred from other regional cancer networks within England.

Eligible patients will receive systemic chemotherapy (in accordance with local protocols) and PIPAC (Doxorubicin 1.5 mg/m2 body surface area Cisplatin 7.5 mg/m2 body surface area). Patients will receive three cycles of systemic chemotherapy interposed with three PIPAC sessions. Chemotherapy cycles will be occur at six weekly intervals.

Following completion of neoadjuvant systemic chemotherapy and PIPAC patients will be restaged. Patients will be considered eligible for D2 radical gastrectomy if the following conditions are met:

(i) negative peritoneal cytology; (ii) absence of macroscopic peritoneal metastasis (PCI 0); (iii) absence of solid organ metastasis (for T4b disease please see point iv below); (iv) expectation of complete (R0) resection of primary tumour; (v) patient considered medically fit for gastrectomy (performance status ≤ 1, absence of organ failure or uncontrolled co-morbidity), and; (vi) provision of informed written consent for treatment (surgery)

Patients who do not meet these criteria will be offered continued palliative and/or best supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma (Tx, Nx) 1,2,3
* Peritoneal cytology +ve or PCI ≤ 3
* No solid organ metastasis 2
* HER2 -ve
* Male/female
* Treatment naïve
* BMI ≥ 18.5 kg/m2 or ≤ 40 kg/m2
* WHO performance status ≤ 1
* Dysphagia score ≤ 2
* Informed written consent

Exclusion Criteria:

* PCI ≥ 4
* Solid organ metastasis
* Positive lymph node disease beyond field of D2 lymphadenectomy
* Peritoneal adhesions precluding complete laparoscopy
* Ascites (greater than trace amount)
* Malignant pleural effusion
* Mechanical bowel obstruction (with the exception of gastric outlet obstruction)
* HER2 +ve
* Patients eligible for immunotherapy
* Uncontrolled co-morbidity
* single/multiple organ failure
* BMI < 18.5 kg/m2 or > 40 kg/m2
* WHO performance status > 1
* Dysphagia score > 2
* Contraindication to chemotherapy
* Pregnancy or breastfeeding
* Haemoglobin <90 g/dL uncorrected with blood transfusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety of combined neoadjuvant systemic chemotherapy and pressurised intraperitoneal aerosol chemotherapy (PIPAC) | 2 years
  Barrier and mitigating factors or the provision of combined neoadjuvant systemic chemotherapy and PIPAC will be assessed. Safety of this intervention in terms of risks to patients and staff will also be evaluated.

SECONDARY OUTCOMES:
Tumour regression | 2 years
  Regression of peritoneal tumour deposits and/or positive peritoneal cytology. Regression will be assesses visually at the time of laparoscopy, by appropriate cross sectional imaging and through histological assessment of acquired samples.
Patient morbidity | 2 years
  Common Toxicity Criteria and Common Terminology Criteria for Adverse Events (Ver. 5) will be used to grade any complications that occur as a consequence of systemic chemotherapy and PIPAC administration. Surgical complications will reported using standard terminologies and graded using the Clavien-Dindo system.
Health related quality of life | 2 years
  Health related quality of life will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) generic questionnaire QLQ-C30 (version 3.0).
Disease recurrence and survival | 5 years
  Peritoneal disease recurrence (assessed by conventional methods), overall and disease-free survival following radical gastrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: George B Hanna, FRCS, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, Hammersmith Hospital Campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No